CLINICAL TRIAL: NCT07316335
Title: The Effect of Cognitive Behavioral Model-Based Psychoeducation on Social Exclusion, Hopelessness, and Relapse Levels in Individuals Diagnosed With Substance Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Seyma Laloglu, specialist nurse, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AİBU-HF-ŞL-01
Record Dates: First submitted 2025-02-25; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Psychoeducation based on cognitive behavioral model; substance use disorder; hope; social exclusion
MeSH Terms: conditions — Substance-Related Disorders; Social Isolation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled experimental type study.44 people planned to be included in the research sample will be selected by simple random method. Then, it was planned to include 22 patients in the experimental group and 22 patients in the control group by randomization method. During this process, a list of 44 patients who voluntarily agreed to participate in the research will be created. In this list, patients will be numbered from 1 to 44. Then, with the software at http://www.randomizer.org, 22 out of 44 numbers will be randomly assigned to the experimental group and 22 to the control group. After the assignment, patients corresponding to the numbers in the experimental group will be included in the experimental group and patients corresponding to the numbers in the control group will be included in the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Before starting the program, the researcher received a Cognitive Behavioral Therapy (CBT) Theoretical Basic Training certificate. During the preparation of the Cognitive Behavioral Model-Based Psychoeducation Program, first of all, studies in the literature and books on the subject were examined, using both domestic and international sources. While creating training topics, the Cognitive Behavioral Model, which includes various cognitive and behavioral approaches designed to achieve the goal at each stage of the relapse process, was used. Each psychoeducation session will focus on planned topics such as informing patients about substance addiction, teaching them how to cope with high-risk situations, providing skills that can prevent relapses, providing impulse management, teaching stress coping skills, and increasing hope. Before starting the application, expert opinions will be presented and arrangements will be made in line with the suggestions.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Theoretical Basic Training Group
- control group (No Intervention): The control group will not be given any training or information during this period. They will continue their normal routines and treatments in daily life. After the training process ends, a post-test will be applied to the control group.
  After the study is completed, psychoeducation will be given to the control group if they request.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) Theoretical Basic Training Group — It was planned to measure the effect of cognitive behavioral model-based psychoeducation on the level of social exclusion and hope in individuals diagnosed with substance use disorder, as well as teaching them to cope with the relapses they struggle with.
  Arms: experimental group

SUMMARY:
This research was planned to measure the effect of cognitive behavioral model-based psychoeducation on the level of social exclusion and hope in individuals diagnosed with substance use disorder, as well as teaching them to cope with the relapses they struggle with.

DETAILED DESCRIPTION:
Substance addiction is a problem that all societies in the world are exposed to and is increasing in society.It is a serious public health problem. Substance use disorder affects individuals despite the negative consequences in bio-psycho-social areas, people continue to use psychoactive substances.a brain that continues with cravings, cravings for substance use, remissions, and relapses is the disease. There are many problems that continue with relapses and vary depending on the individual's addiction process. In the treatment of problematic substance use disorders, in addition to pharmacological treatment, psychotherapy and psychosocial approaches in which the person can actively participate Adding it to the treatment increases the success rate of the treatment. Psychosocial in substance addiction cognitive behavioral model-based approach, one of the intervention programs, It appears as one of the preferred intervention programs for addicts. Relapse prevention based on cognitive behavioral foundations developed by Marlatt and Gordon relapse prevention program helps reduce the risk of relapse in conditions such as substance use disorders focuses. This program includes various cognitive-behavioral skills that can be effective at different stages of the process. includes approaches. These approaches aim to increase individuals' hopes and improve their social skills.

It aims to develop and strengthen skills in coping with high-risk situationsProgram, It includes strategies that will help individuals regain their self-confidence. This, to ensure that individuals do not despair during the recovery process and that their motivation remains high.

supports their retention. Individuals are healthier and more effective in social interactions and relationships.

aims to communicate. Developing social skills as well as strengthening support systems It also focuses on supporting positive social interactions. The program allows individuals to It offers strategies to help students cope with high-risk situations associated with their use. This skills to cope with situations, the risk of falling behind when faced with risky situations, can reduce it. This relapse prevention program enables individuals to achieve sustainable improvement throughout the treatment process. While helping them achieve their goals, it also aims to minimize the risk of falling behind.

Integration of cognitive behavioral approaches, individuals' healthy lifestyle choices It supports them to become aware of and strengthen these choicesIn this way, they are more likely to learn to cope with and sustain chronic conditions such as substance use disorders.

becomes.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18 and 65,
2. Being diagnosed with substance use disorder according to DSM-V,
3. Absence of comorbid diagnosis (bipolar disorder, anorexia/bulimia nervosa, psychotic symptoms)

Exclusion Criteria:

1. People experiencing acute exacerbations
2. People who continue to use alcohol or substances

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
implementation of psychoeducation based on the cognitive behavioral model - Social Exclusion Level | 16 weeks
  Outcome Measure: Social Exclusion Scale
  Description:
  The Social Exclusion Scale will be used to assess participants' levels of exclusion from social relationships and withdrawal from social participation. Total scale scores will be used for quantitative analysis. The minimum and maximum possible scores and the interpretation of higher scores (indicating greater or lower levels of social exclusion) will be specified in the data analysis plan.
implementation of psychoeducation based on the cognitive behavioral model - Hopelessness Level | 16 weeks
  Outcome Measure: Beck Hopelessness Scale (BHS)
  Description:
  The Beck Hopelessness Scale will be used to measure participants' levels of hopelessness. Total scores obtained from the scale will reflect the severity of hopelessness. The minimum and maximum possible scores and the interpretation that higher scores indicate higher levels of hopelessness

SECONDARY OUTCOMES:
Relapse Coping Skills Scale | 8 weeks
  1. Relapse Coping Level
  Outcome Measure: Relapse Coping Skills Scale
  Description:
  Participants' levels of coping with relapse will be assessed using a structured scale or subscale designed to evaluate relapse coping skills. Total scores obtained from the scale will be used to reflect participants' levels of relapse coping. The score range and interpretation of higher scores will be specified in the data analysis plan.
Substance Use Coping Strategies Scale | 8 weeks
  2. Substance Use Coping Strategies
  Outcome Measure: Substance Use Coping Strategies Scale
  Description:
  Coping strategies related to substance use will be assessed using a psychometric scale measuring cognitive and behavioral coping skills. Outcomes will be analyzed based on total scale scores, reflecting participants' use of adaptive coping strategies.